CLINICAL TRIAL: NCT02813655
Title: Evaluation of the Effectiveness and Tolerance of Tetracosactide Synacthen® in the Treatment of Post Dural Puncture Headaches (ESYBRECHE)
Acronym: ESYBRECHE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis and decision of the independent committee, investigators and sponsor (futility) (2023/10/05)
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 69HCL15_0429; 2015-003357-17 (EudraCT Number)
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Post-dural Puncture Headache
Keywords: tetracosactide; Synacthène®; cosyntropin; post-dural syndrom; post-dural puncture headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Cosyntropin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): Tetracosactide (Synacthène®)
  Interventions: Drug: Tetracosactide (Synacthène®)
- Control arm (Placebo Comparator): placebo saline (0.9% NaCl)
  Interventions: Drug: placebo saline (0.9% NaCl)

INTERVENTIONS:
Drug: Tetracosactide (Synacthène®) — Tetracosactide, manufactured by Sigma-Tau® laboratories and marketed under the name of Synacthène®.
  All women who received epidural or combined spinal-epidural labour analgesia and presenting post-partum post dural puncture headache were randomized. The patient will receive 1 mg of Synacthène® intravenously during 20 minutes. Four vials of 1 ml of Synacthène® will be added to a bag of 100 ml of physiological saline. The injection of study treatment must be done within 6 hours after the inclusion. Monitoring of the patient is carried out throughout the duration of administration of the drug, then between H2 and H6, D1, D2, D3 and D15.
  Arms: Experimental arm
Drug: placebo saline (0.9% NaCl) — placebo saline manufactured by the laboratory Aguettant: 10ml vial, 4 mL will be collected and added to a bag of 100 ml of saline.
  All women who received epidural or combined spinal-epidural labour analgesia and presenting post-partum post dural puncture headache were randomized. The patient will receive 4 ml of placebo saline added to a bag of 100 ml of physiological saline ( 104 ml of physiological saline). The injection of study treatment must be done within 6 hours after the inclusion. Monitoring of the patient is carried out throughout the duration of administration of the drug, then between H2 and H6, D1, D2, D3 and D15.
  Arms: Control arm

SUMMARY:
The aim of the study is to assess the efficacy and safety of Synacthène® versus placebo in the treatment of post-dural puncture syndrome in patients receiving epidural analgesia, spinal analgesia, or combined spinal-epidural analgesia for labour.

ELIGIBILITY:
Inclusion Criteria:

All women who received epidural, spinal, or combined spinal-epidural labour analgesia and presenting post-dural puncture headache:

* Intense: with ≥3 / 10 numerical rating pain scale
* Appearing within 5 days after delivery
* Aggravating in sitting or standing position and / or improving supine
* Can be associated with one of the following criteria: tinnitus, nausea, photophobia, neck stiffness or pain, hearing loss
* After exclusion of clinically differential diagnoses (preeclampsia or eclampsia, cerebral venous thrombosis, migraine)
* Age greater than or equal to 18 years
* Affiliation to social security scheme
* Inform Consent signed after oral and written information

Exclusion Criteria:

* Presence of diplopia (indication of immediate blood patch)
* Contraindication to ACTH or Synacthène® (unbalanced hypertension, uncontrolled diabetes, uncontrolled psychosis, infectious viral disease state or evolving)
* Processing of Torsade de Pointe provider (astenizole, bepridil, erythromycin IV, halofantrine, pentamidine, sparfloxacin, sultopride, terfenadine, vincamine)
* Live vaccine in the months prior to inclusion
* Hypersensitivity to Synacthène®
* Patient who have previously received Synacthène® after delivery
* Contraindication to blood patch (fever or leukocytosis, HIV or HCV patient)
* Eclampsia or preeclampsia during this pregnancy
* Patient who have received prophylactic blood patch (at diagnosis of Accidental Dural Puncture)
* Minor under 18 or protected
* Psychological disorders do not allowing informed consent
* Refusal of participation in the study or participation in another ongoing interventional study
* Withdrawal of consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Rate of blood patch use | Day 15
  Assessment of the rate of blood patch use between experimental group (Synacthène®) and control group between day 0 and day 15.

SECONDARY OUTCOMES:
Side effects | Day 15
  Type, severity and number of side effects in each group (control and experimental) between day 0 and day 15
Duration of headache | Day 15
  Duration of headache in each group (control and experimental) between day 0 and day 15
Intensity of headache | Day 15
  Intensity of headache in each group (control and experimental) between day 0 and day 15
analgesic use (type and duration) in each group (control and experimental) | Day 15
  analgesic use (type and duration) in each group (control and experimental) between day 0 and day 15
blood-patch number | Day 15
  blood-patch number per patient in each group (control and experimental) between day 0 and day 15
Time to first analgesic use after injection of treatment (Synacthène® or placebo) | Day 15

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron
  - Hospices Civils de Lyon / hôpital de la Croix rousse, Lyon

REFERENCES:
- [Result] Dziadzko M, Bouvet L, Steer N, Depaulis C, Pradat P, Joubert F, Lalande L, Chassard D, Aubrun F. No effect of tetracosactide for treatment of postdural puncture headaches in parturient women: a double-blind randomised controlled clinical trial. Br J Anaesth. 2025 Jul;135(1):148-154. doi: 10.1016/j.bja.2025.04.012. Epub 2025 May 19. PMID 40393818
- [Derived] Depaulis C, Steer N, Garessus L, Chassard D, Aubrun F. Evaluation of the effectiveness and tolerance of tetracosactide in the treatment of post-dural puncture headaches (ESYBRECHE): a study protocol for a randomised controlled trial. Trials. 2020 Jan 8;21(1):55. doi: 10.1186/s13063-019-4015-y. PMID 31915040